CLINICAL TRIAL: NCT00440570
Title: Treatment of Advanced Cancer With Amplitude-modulated Electromagnetic Fields of Low Intensity by Means of an Intrabuccal Probe
Brief Title: A Study of Therapeutic Amplitude-modulated Electromagnetic Fields in Advanced Tumors
Acronym: THBC001
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pasche, Boris, M.D. (Individual)
Collaborators: Barbault, Alexandre, M.S. (Individual)
Responsible Party: Boris Pasche, Boris Pasche
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 001
Record Dates: First submitted 2007-02-24; First posted 2007-02-27 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Cancer; Brain Tumor
Keywords: cancer; electromagnetic fields; treatment
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Low levels of amplitude-modulated electromagnetic fields
Device: Emitter of low levels of amplitude-modulated electromagnetic fields

SUMMARY:
In vitro studies suggest that low levels of amplitude-modulated electromagnetic fields may modify cell growth. We have identified specific frequencies that may block cancer cell growth. We have developed a device delivering low levels of amplitude-modulated electromagnetic fields. The device is connected to a spoon-like coupler, which is placed in the patient's mouth during treatment. We will conduct a feasibility study consisting of three daily ambulatory treatments until disease progression.

DETAILED DESCRIPTION:
Background: In vitro studies suggest that low levels of amplitude-modulated electromagnetic fields may modify cell growth. We have identified specific frequencies that may block cancer cell growth. We have developed a portable and programmable device delivering low levels of amplitude-modulated electromagnetic fields. The device is connected to a spoon-like coupler, which is placed in the patient's mouth during treatment.

Methods: We will conducted a feasibility study consisting of three daily treatments. All patients with advanced solid tumors and measurable disease will be eligible, irrespective of prior treatments. Patients will be assessed with laboratory exams (complete blood count, comprehensive profile, tumor markers), imaging studies every other month for the first six months, every third month thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Advanced tumor that is either metastatic or inoperable

Exclusion Criteria:

* Pregnancy,
* Other simultaneous anticancer therapies,
* ECOG performance status less than 3

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2
Dates: Start 2004-10; Primary Completion 2006-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety of daily administration of amplitude-modulated electromagnetic fields in patients with advanced cancer

SECONDARY OUTCOMES:
Complete blood count, comprehensive chemistry profile, tumor markers
Tumor assessment as per RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Boris C Pasche, MD, PhD, Principal Investigator — Cabinet Médical Avenue de la gare 6
Locations (1):
- Cabinet Médical Avenue de la gare 6, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Barbault A, Costa FP, Bottger B, Munden RF, Bomholt F, Kuster N, Pasche B. Amplitude-modulated electromagnetic fields for the treatment of cancer: discovery of tumor-specific frequencies and assessment of a novel therapeutic approach. J Exp Clin Cancer Res. 2009 Apr 14;28(1):51. doi: 10.1186/1756-9966-28-51. PMID 19366446